CLINICAL TRIAL: NCT00343083
Title: A Phase II Study of Evaluation of Cetuximab (ERBITUX) and Concurrent Carboplatin, Paclitaxel & Radiotherapy in the Management of Patients With Advanced Locoregional Squamous Cell Carcinomas of the Head and Neck
Brief Title: Evaluation of Cetuximab (ERBITUX) and Concurrent Carboplatin, Paclitaxel & Radiotherapy in the Management of Patients With Advanced Locoregional Squamous Cell Carcinomas of the Head and Neck (GCC 0442)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00042712; CA225092
Record Dates: First submitted 2006-06-20; First posted 2006-06-22 (Estimated); Results first posted 2014-04-09 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Cancer of Head and Neck
Keywords: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab; Paclitaxel; Carboplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab comparison for Head and Neck Cancer (Experimental): To report the mature data of a prospective Phase II trial designed to evaluate the efficacy of an epidermal growth factor receptor inhibitor cetuximab (CTX) added to the concurrent therapy of weekly paclitaxel/carboplatin (PC) and daily radiation therapy (RT).
  Both chemotherapy and radiation will be given on a weekly basis (see interventions for details).
  Interventions: Drug: Erbitux, Paclitaxel & Carboplatin; Radiation: Radiation

INTERVENTIONS:
Drug: Erbitux, Paclitaxel & Carboplatin — Paclitaxel, 40 mg/m2/week,
  1-hour infusion (weeks 2-9.Paclitaxel will be administered on a weekly schedule at a dose of 40mg/m2 IV by 1-hour infusion prior to cetuximab dose.
  Cetuximab: 400 mg/m2 IV (initial dose) week 1 then 250 mg/m2 IV weekly for 8 weeks weeks 2-9). Cetuximab will be administered 400mg/m2 IV on Day 1, then the first 250 mg/m2 IV dose will be given on day 8 (week 2) prior to carboplatin dose.
  Carboplatin, AUC=2/week as a 30 minute infusion after cetuximab infusion (weeks 2-9)Carboplatin will be administered at a dose of AUC = 2/week IV bolus each week and will be administered prior to head and neck irradiation dose. (Carboplatin: AUC=2/week x 8 weeks (weeks 2-9)
  Other Names: Taxol, Erbitux
Radiation: Radiation — XRT=Radiotherapy 1.8 Gy radiation/day, 5 days a week for a total of 70.2 Gy.(weeks 2-9) - IMRT is allowed

SUMMARY:
The purpose of this study is to evaluate the response of the tumor to the treatment regimen that will be used in this study. This study will also test the safety of cetuximab (C225), given with chemotherapy and radiation therapy. We also want to see what effects (good and bad) cetuximab, chemotherapy, and radiation therapy have head & neck cancer.

C225 has been designed to stop the growth of the tumor by blocking certain chemical pathways that lead to tumor cell growth. In prior studies with head & neck cancer patients, C225 has delayed tumor growth and provided relief of symptoms in some patients.

DETAILED DESCRIPTION:
Primary Objective- To evaluate whether the addition of Cetuximab (C225) in combination with chemotherapy and radiation can cause an enhanced anti-tumor effect resulting in improving local regional control of patients with locally advanced, unresectable squamous cell carcinoma of head and neck. (SCCHN).

OVERVIEW OF STUDY DESIGN Open label, non-randomized, single arm trial.

P = Paclitaxel will be administered on a weekly schedule at a dose of 40mg/m2 IV by 1-hour infusion prior to cetuximab dose. This will be administered for a total of 8 weeks (from weeks 2-9)

C225 = Cetuximab: 400 mg/m2 IV will be given as the initial OR loading dose in week 1 and then 250 mg/m2 IV weekly will be given for 8 weeks (weeks 2-9).

C = Carboplatin will be given at a dose of AUC=2/week - will be administered as a 30 minute infusion after cetuximab infusion (weeks 2-9)

RT = Radiation therapy will be delivered at 1.8 Gy fraction/day, 5 days a week for a total of 70.2 Gy. RT will be given from weeks 2-9.

Note: Sequence of administration will be paclitaxel followed by cetuximab followed by carboplatin followed by XRT.

Approximately 60 patients from MSGCC/BVAMC will participate in this study. Prior to entering the study the doctor will examine the patient and order blood tests ( which will be done by blood draw, approximately 2 tablespoons) and tests to measure the patients disease (scans). The patient will also be evaluated by a dietician who will follow the patient throughout the course of the therapy to help the patient meet his/her nutritional needs

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proved locally advanced squamous cell carcinoma of the head and neck of all primary sites. The following TNM stages by sites will be eligible.Oral cavity, Pharynx, Larynx, Nasopharynx, paranasal sinuses, Oral cavity, Pharynx, Larynx, Nasopharynx, paranasal sinuses- T4 N0 N1 N2-A,B,C N3, T3 N0 N1 N2-A,B,C N3 Any T N2-A,B,C N3 Unknown primary Tx N2-A,B,C N3 Note: Only clearly unresectable T4 N0 lesions are eligible for study provided the reasons for unresectability are due to extensive anatomic involvement and are outlined by the surgeon
2. Patients must have signed an approved informed consent.
3. Patients with Performance Status 0-2.
4. No evidence of distant metastatic disease.
5. No previous radiation therapy.
6. No previous chemotherapy.
7. Patients must be greater than 18 years of age.
8. Women of child bearing potential (WOCBP) must have a negative pregnancy test within 7 days of treatment. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
9. Pretreatment evaluations include:

   History and physical examination within four weeks prior to study entry Dental evaluation Medical oncology examination to evaluate medical contraindications prior to start of chemotherapy
10. Adequate renal & bone marrow function determined by the following laboratory parameters:

    ANC greater than or equal to 1500/mm3; platelets greater than or equal to 100,000/mm3; hemoglobin greater than or equal to 8.0 g/dl; Serum Creatinine less than or equal to 2.0 mg/dl, Total bilirubin less than 1.5 X the ULIN; AST/ALT less than 3 times the ULN, Creatinine Clearance greater than or equal to 50 cc/min
11. Evidence of measurable disease.
12. No evidence of concomitant malignancy except for non-melanomatous skin cancer (controlled or controllable) or carcinoma in situ of the cervix.

Exclusion Criteria:

Any of the following criteria will make the patient ineligible to participate in this study:

1. Acute hepatitis or known HIV.
2. Active or uncontrolled infection.
3. Significant history of concomitant life threatening / uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and known cardiomyopathy with decreased ejection fraction, cardiac arrhythmia
4. Prior therapy which specifically and directly targets the EGFR pathway.
5. Prior severe infusion reaction to a monoclonal antibody.
6. Any concurrent chemotherapy not indicated in the study protocol or any other investigational agent(s).
7. Women of childbearing potential (WOCBP) and male participants who are unwilling or unable to use an effective method to avoid pregnancy for the entire study period
8. Preexisting clinically significant neuropathy.
9. Patients with loco-regional recurrences from any site with no prior radiation therapy and not amenable for salvage surgery are not eligible for study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-12; Primary Completion 2011-06 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Suntharalingam, M.D, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland & Baltimore VA medical centre, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cetuximab (ERBITUX) and Concurrent Carboplatin: . Radiation will be given at a dose of 1.8 Gy. for a total of 70.2 Gy. Chemotherapy will be given every week for a total of 8 weeks. Paclitaxel will be given at a dose of 40 mg/m2 as a 1 hour infusion dose followed by cetuximab and then carboplatin AUC = 2/week.
  The initial dose of cetuximab is 400 mg/m2 IV on day 1, followed by weekly infusions at 250 mg/m2 IV.
Period: Overall Study
Arm/Group | Cetuximab (ERBITUX) and Concurrent Carboplatin
Started | 43
Completed | 22
Not Completed | 21

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab (ERBITUX) and Concurrent Carboplatin
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is the Local Regional Control Rate Assessed 3 Months Post Completion of Radiation Therapy.
Description: The local regional control rate was assessed 3 months post completion of radiation therapy based on either MRI or CT and clinical exam.
Time Frame: 3 months
Measure: Number; unit: participants
Groups:
- Concurrent Chemo Raditaion Wtih Cetuximab: The addition of CTX to weekly PC and daily RT.
Arm/Group | Concurrent Chemo Raditaion Wtih Cetuximab
Number analyzed (Participants) | 43
participants | 43

2. Secondary Outcome: Local Regional Control at 2 Years
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Concurrent Chemo Raditaion Wtih Cetuximab
Number analyzed (Participants) | 43
percentage of participants | 72 (38)

3. Secondary Outcome: Overall Survival and Disease-free Survival
Time Frame: 3 years (overall) 2 years disease-free
Measure: Number; unit: percentage of participants
Arm/Group | Concurrent Chemo Raditaion Wtih Cetuximab
Number analyzed (Participants) | 43
percentage of participants
  overall survival | 59 (38)
  disease-free survival | 58

4. Secondary Outcome: Pathological Response to Cetuximab
Description: Adding CTX to weekly PC and daily RT. CBC and Chemistry panel blood testing
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Concurrent Chemo Raditaion Wtih Cetuximab
Number analyzed (Participants) | 43
participants | 43

5. Secondary Outcome: Percentage of Participants With Grade 3 Toxicities of Cetuximab
Description: One of the more serious side effects of cetuximab therapy is the incidence of acne-like rash. This rash rarely leads to dose reductions or termination of therapy. It is generally reversible.
  Further severe infusion reactions include but are not limited to: fevers, chills, rigors, urticaria, pruritis, rash, hypotension, N/V, HA, bronchospasm, dyspnea, wheezing, angioedema, dizziness, anaphylaxis, and cardiac arrest. Therefore, pretreatment with diphenhydramine 30-60 min. before administration is standard of care. Other common side effects include photosensitivity, hypomagnesemia due to magnesium wasting, and less commonly pulmonary and cardiac toxicity.
Time Frame: 9 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Concurrent Chemo Raditaion Wtih Cetuximab
Number analyzed (Participants) | 43
percentage of participants
  mucositis | 79 (43)
  rash | 9
  leukopenia | 19
  neutropenia | 19
  RT dermatisis | 16

6. Secondary Outcome: Clinical Complete Response Rate of This Regimen in the Population
Description: What is the the complete response (CR) rate at the completion of therapy.
Time Frame: 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Concurrent Chemo Raditaion Wtih Cetuximab
Number analyzed (Participants) | 43
percentage of participants | 84 (38)

ADVERSE EVENTS:
Arm/Group | Cetuximab (ERBITUX) and Concurrent Carboplatin
Serious Adverse Events (participants affected / at risk) | 3/43
Other Adverse Events (participants affected / at risk) | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab (ERBITUX) and Concurrent Carboplatin (N=43)
Anaphylactic reaction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) — 3 patients developed a Grade IV anaphylactic reaction to the loading dose of Erbitux (week 1) and were taken off protocol hence withdrawn due to toxicity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No